CLINICAL TRIAL: NCT01244139
Title: A Randomized, Blinded, Placebo-Controlled, Serial-Cohort, Multiple Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of BIIB033 in Subjects With Multiple Sclerosis
Brief Title: Safety Study of BIIB033 in Subjects With Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple
Other Study IDs: 215MS101
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Relapsing-Remitting Multiple Sclerosis; Multiple Sclerosis
Keywords: BIIB033; Multiple Sclerosis; anti-LINGO-1 antibody; Relapsing Remitting MS; remyelination; myelin repair; Multiple ascending dose; Secondary progessive MS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — opicinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active study drug (Experimental): Treatment
  Interventions: Drug: BIIB033
- Comparator (Experimental): Dummy drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB033 — IV infusion of 0.3, 1, 3, 10, 30, 60 or 100 mg/kg
  Arms: Active study drug
Drug: Placebo — IV infusion dummy drug
  Arms: Comparator

SUMMARY:
The main purpose of the study is to evaluate the safety, tolerability, and pharmacokinetic profile of two intravenous infusions of BIIB033 administered two weeks apart in subjects with MS.

Approximately 42 MS subjects are planned to be enrolled in the study in 7 separate groups (i.e., 6 subjects per group). Each subsequent group will be administered a higher dose of BIIB033. Before a higher dose group is allowed to start, a Drug Safety Review Committee will review all safety data from previous groups enrolled, as well as data from another study where BIIB033 is being administered to healthy volunteers (215HV101).

DETAILED DESCRIPTION:
BIIB033 is a protein that acts on certain types of brain cells by blocking the function of another protein called LINGO-1. It is believed that LINGO-1 is one of the reasons why nerves in the brain of patients with MS do not repair well. It is thought BIIB033 may improve MS by repairing damaged nerve tissue. LINGO-1 is also present in the brain of healthy people.

Subjects will take part in the 215MS101 study for up to 28 weeks. This includes a 4-week screening period, a 2 week treatment period in which 2 doses of BIIB033 are given, and a post-dosing safety follow up period of up to 22 weeks (depending on dose cohort).

The study tests vary at each of the individual visits and may include:

medical history evaluation, height and weight assessment, physical examination, neurological examination, vital signs assessment (pulse, respiratory rate, blood pressure, and temperature), MS performance score, electrocardiogram, cardiac monitoring, routine blood and urine tests, drug concentration testing of the blood, hepatitis and HIV tests, blood clotting tests, brain MRI scan, lumbar puncture, and drugs of abuse screen and pregnancy test.

ELIGIBILITY:
Inclusion Criteria:

* Give informed consnet
* Aged 18 to 60 years
* Have relapsing remitting MS or secondary progressive MS
* EDSS score of 1 to 6 inclusive
* Body mass index of 18 to 30 kg/m2
* Commitment to use effective contraception 6 months after last dose of study drug Treatment with any interferon beta or glatiramer acetate is allowed to continue during the study as long as the initiation of treatment was at least 3 months and the dose is stable.

Key Exclusion Criteria:

* Primary progressive MS
* Any significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, allergic or anaphylactic reactions or other major disease
* Clinically significant lab value at screening outside of normal range
* Clinically significant ECG abnormality
* Contraindication to MRI scans or lumbar punctures
* Plans to undergo elective surgery during study
* An MS relapse that has not resolved within 30 days before screening
* History or postive test result for Hepatitis B, C and HIV
* Serious infections within 3 months prior to Day -1
* Treatment with MS medication within 12 months prior to Day -1: natalizumab, daclizumab, azathioprine, methotrexate, iV immunoglobulin, plasmapheresis or mycophenolate motefil
* Prior treatment with total lymphoid irradiation, T cell or T-cell receptor vaccination, alemtuzumab, mitoxantone, cyclophosphamide, rituximab, fingolimod.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and tolerability profile of two IV infusions of BIIB033 in subjects with MS | For duration of study / 6 months
Identify incidence and types of adverse events | For duration of study / 6 months
The incidence of serious adverse events | For duration of study / 6 months
Changes from baseline in clinical lab assessments and vital signs | For duration of study / 6 months
Changes form baseline in other safety measures: physical and neurological examinations, brain MRIs, and ECGs | For duration of study / 6 months

SECONDARY OUTCOMES:
Assess the repeat-dose serum PK profile of BIIB033 | For duration of study / 6 months
Assess the repeat-dose immunogenicity of BIIB033 | For duration of study / 6 months
Measure the concentration of BIIB033 in the cerebrospinal fluid | At specified timepoints in the study
Explore potential biomarkers of BIIB033 activity in the periphery and in the central nervous system | At specified timepoints in the study

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Centennial, Colorado, United States

REFERENCES:
- [Background] Tran JQ, Rana J, Barkhof F, Melamed I, Gevorkyan H, Wattjes MP, de Jong R, Brosofsky K, Ray S, Xu L, Zhao J, Parr E, Cadavid D. Randomized phase I trials of the safety/tolerability of anti-LINGO-1 monoclonal antibody BIIB033. Neurol Neuroimmunol Neuroinflamm. 2014 Aug 21;1(2):e18. doi: 10.1212/NXI.0000000000000018. eCollection 2014 Aug. PMID 25340070
- [Derived] Boyd A, Zhang H, Williams A. Insufficient OPC migration into demyelinated lesions is a cause of poor remyelination in MS and mouse models. Acta Neuropathol. 2013 Jun;125(6):841-59. doi: 10.1007/s00401-013-1112-y. Epub 2013 Apr 18. PMID 23595275